CLINICAL TRIAL: NCT04711616
Title: Physical Therapy Interventions Following Arthroscopic Rotator Cuff Repair: A Prospective Single Group Interventional Study
Brief Title: Physical Therapy Interventions Following Arthroscopic Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Hyun-Joong Kim, Principal Investigator, Sahmyook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2-1040781-A-N-012021012HR
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Rotator Cuff Injuries; Pain, Postoperative; Kinesiophobia
MeSH Terms: conditions — Rotator Cuff Injuries; Pain, Postoperative; Kinesiophobia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- physical therapy intervention (Experimental)
  Interventions: Behavioral: physical therapy intervention

INTERVENTIONS:
Behavioral: physical therapy intervention — physical therapy interventions include thermal therapy, electrical therapy, manual therapy, and therapeutic exercise.

SUMMARY:
In the post-arthroscopic rotator cuff repair (ARCR) management, physical therapy intervention is an important factor in bringing about a clinically positive prognosis. However, no conclusive therapeutic evidence has been found for various physical therapy interventions. In this study, the investigators would like to investigate the effects of physical therapy interventions on ARCR patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years old
* In case of 2 weeks after receiving arthroscopic rotator cuff repair
* When the participants wishes to enroll in the study

Exclusion Criteria:

* 65 years old or older
* If the tear area is large and augmentation is performed
* If there is a previous surgical history at the surgical site
* Osteoarthritis in the shoulder joint

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Change from baseline pain intensity at 12 weeks
  A numeric pain rating scale (NPRS) consisting of 11 points in total from 0 points (no pain) to 10 points (the most severe pain imaginable) is used. The lower the score, the less the pain.

CONTACTS AND LOCATIONS:
Locations (1):
- The Better Hospital, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: Yes